CLINICAL TRIAL: NCT00087906
Title: Disability and Health Outcomes in COPD
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1262; R01HL077618 (NIH)
Record Dates: First submitted 2004-07-15; First posted 2004-07-19 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Obstructive Pulmonary Disease; Lung Diseases
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To test a conceptual model of how disability develops in chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
BACKGROUND:

Background. COPD is a common chronic health condition. Because current medical treatments have minimal impact on disease progression, a strategy to prevent COPD-related disability would have important clinical and public health benefits.

DESIGN NARRATIVE:

The study will test a specific conceptual model of how disability develops in COPD. The aims are: (1) To evaluate the impact of respiratory impairment, especially pulmonary function impairment, on the risk of functional limitation in COPD. Using a control group, to elucidate the prevalence of respiratory impairment, functional limitation, and disability that is directly attributable to COPD. (2) In adults with COPD, to delineate the longitudinal effect of functional limitation on the risk of incident disability. The investigators hypothesize that development of functional limitation, and not pulmonary function impairment, is the major determinant of disability. (3) To determine the prospective impact of disability on the risk of future adverse health outcomes. The investigators will assemble a prospective cohort of 1200 randomly sampled adults with COPD who are members of a large regional health maintenance organization. A matched control group of 300 subjects will be recruited. Subjects will undergo a detailed physical assessment that measures respiratory impairment (e.g., pulmonary function) and functional limitation (e.g., lower extremity function, muscle strength, exercise performance, and cognitive function). Structured telephone interviews will ascertain disability outcomes at baseline and 18-month prospective follow-up. The investigators will also study the modulating effects of specific risk factors and protective factors on the progression from functional limitation to COPD-related disability, including psychological factors, environmental exposures, and health care process factors.

ELIGIBILITY:
Inclusion:

1. COPD diagnosis and
2. Medication use for cases

Exclusion:

1. Withdrew from Kaiser Plan prior to baseline contact

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: We recruited persons with COPD for what we came to term the "FLOW study." The original project was funded to complete two interviews and a single research clinic evaluation. In addition to completing this original program of work successfully, we also carried out follow-up research clinic visits for 667 subjects. These supplemental examinations were made possible through research funding support from the Flight Attendants Medical Research Foundation (FAMRI).
Sampling Method: Probability Sample
Enrollment: 1589 (Actual)
Dates: Start 2004-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
COPD Disability | 10 years
  Observational self-reported impairment in valued life activities.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Blanc, MD, Principal Investigator — University of California at San Francisco

IPD SHARING:
Plan to Share IPD: No